CLINICAL TRIAL: NCT02973009
Title: Impact of the Systematic Closure of the Epigastric Trocar on Postoperative Incisional Hernia After Sleeve Gastrectomy Rate of First Intention. Monocentric Study, Before / After Prospective.
Acronym: TROCSLEEVE
Status: Withdrawn | Type: Observational
Why Stopped: investigator choice
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2016_843_0031
Record Dates: First submitted 2016-11-14; First posted 2016-11-25 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Bariatric Surgery
Keywords: The Sleeve Gastrectomy (SG); bariatric surgery; laparoscopy; systematic closure of the epigastric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The Sleeve Gastrectomy (SG) is a bariatric surgery procedure performed by laparoscopic booming in recent years.

This is an effective intervention on weight loss over the long term with few early postoperative complications and low morbidity in the long term.

Obesity is considered as a risk factor for hernia full after surgery by laparoscopy with a relative risk of 29% in connection with cholecystectomy.

Several series showed a rupture rate on trocar from 0 to 0.7%, but each time with a clinical evaluation.

Recently, it was shown eventrations rate between 26 and 38% under the Roux-en-Y gastric bypass with a rupture rate increased on epigastric trocar. The assessment in the context of this series was ultrasound.

Recent data suggest that the absence of closure of the epigastric trocar of 12mm through an SG of first intention was associated with a hernia rate of 17% with a scannographic evaluation.

Also, recently, Tabone suggests that the systematic closure of the epigastric trocar site would not be as effective as lateralize inserting the trocar from the white line of the abdomen. Change the positioning of this trocar induce an additional difficulty in handling instruments for the realization of the SG with an désaxassion instruments, a conflict between the instruments for the realization of the SG and the optical laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* major patients (≥ 18 years) who underwent SG 1st intention by laparoscopy as part of the surgical management of obesity.

Exclusion Criteria:

* antecedent of previous gastric band.
* History of SG (repeat-SG).
* median laparotomy history or subcostal right.
* SG performed as an ambulatory surgery.
* Patients with early postoperative complications (≤ J90) specific to the SG (postoperative gastric fistula, postoperative bleeding, hematoma or postoperative intra-abdominal abscess)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: major patients who underwent SG 1st intention by laparoscopy as part of the surgical management of obesity
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2017-05-16 (Actual); Study Completion 2017-05-16 (Actual)

PRIMARY OUTCOMES:
systematic closure of the epigastric trocar | 1 year
  Test the hypothesis that the systematic closure of the epigastric trocar 12 mm would reduce by three the number of rupture on epigastric trocar after SG first intent

SECONDARY OUTCOMES:
rate of incisional hernia. | 1 year
  Evaluate the rate of incisional hernia at 1 year after 1st SG intention.
rate of rupture opposite | 1 year
  To evaluate the rate of rupture opposite the closure of the open laparoscopy incision closed using the conventional technique (Deguines JB, Qassemyar Q Dhahri A Brehant O, Fuks D Verhaeghe P Regimbeau JM. Technique of open laparoscopy .. for supramesocolic surgery in obese patients Surg Endosc 2010 Aug; 24 (8): 2053-5) from the rupture rate over the epigastric port with the use of WECK EFx ™ (Teleflex Medical SAS, F-31460 the Faget, France).
Morbidity | 1 year
  Morbidity related to the closing act of the epigastric trocar (organ wound, local hematoma, surgical site infection).
duration of the closure of the epigastric trocar. | during surgery
  Evaluation of the duration of the closure of the epigastric trocar.
duration of the implementation of the device | 1 year
  Analysis of the evolution of the duration of the implementation of the device

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc REGIMBEAU, professor, Principal Investigator — CHU amiens-Picardie